CLINICAL TRIAL: NCT02457936
Title: Examining Cognitive Mechanisms of Clinical Improvement Following Mindfulness Based Cognitive Therapy for Depressed Individuals
Brief Title: Examining Cognitive Mechanisms of Clinical Improvement Following Mindfulness Based Therapy for Depressed Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jonathan Greenberg, Postdoctoral research fellow, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P002481; K23AT010653-01A1 (NIH)
Record Dates: First submitted 2015-05-20; First posted 2015-05-29 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2017-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (MBCT) (Experimental): This group will receive 8 weeks of Mindfulness Based Cognitive Therapy
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Waiting list (Active Comparator): This group will be tested twice 8-10 weeks apart and then receive 8 weeks of Mindfulness Based Cognitive Therapy
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — 8 weekly meetings in which basic mindfulness and meditation skills are taught, such as breathing meditation, body scan meditation, open awareness meditation, movement meditation, and targeting depression related cognitions and emotions in a mindful manner, as well as awareness exercises, group discussions, and daily home meditation practice routines

SUMMARY:
Depression one of the leading causes of disability worldwide. Individuals suffering from depression typically exhibit impairments in various mental abilities, such as the ability to effectively direct and control attention and the ability to switch between thinking about different things and concepts (commonly referred to as "cognitive flexibility").

Mindfulness meditation training is a technique which involves focusing one's awareness on the present moment, while calmly acknowledging and accepting one's feelings, thoughts, and bodily sensations. It has been well documented to improve depressive symptoms and prevent recurrence of depressive episodes, yet little is known about how mindfulness does so and what are the underlying mental mechanisms involved. Here the investigators propose to examine the efficacy of an 8-week mindfulness training program in improving the ability to direct and control attention, as well as in cognitive flexibility.

Individuals diagnosed with recurrent depression will undergo an 8-week mindfulness training program. Participants' depressive symptoms as well as their performance on measures of attention and cognitive flexibility will be examined. Participants will be assigned to mindfulness training or a wait-list control group. Half of the participants will be examined before and after the mindfulness training program and the other half will be tested 8-weeks apart and then begin their training.

ELIGIBILITY:
Inclusion Criteria:

* Reporting dysphoria for at least two months prior
* HAM-D score of at least 11
* No history of psychiatric disorders of psychotic features, neurological disorders, or substance abuse in the past 6 months
* Verified age between 18-65 years old
* Had no suicidal attempts during the past six months
* No prior experience with MBCT or other systematic meditation programs

Exclusion Criteria:

* History of psychosis, neurological disorder, and substance abuse for the past 6 months
* Suicide attempt in past 6 months
* Prior experience with MBCT or other systematic meditation program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms as measured by the Hamilton Depression Rating Scale | Once upon recruitment (baseline), and a second time at 8-10 weeks following the MBCT program
Change from baseline in cognitive flexibility, as measured by a computer task involving task-switching and by the Torrance Test for Creative Thinking | Once upon recruitment (baseline), and a second time at 8-10 weeks following the MBCT program
Change from baseline in attention regulation, as measured by the Attention Network Test | Once upon recruitment (baseline), and a second time at 8-10 weeks following the MBCT program

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Greenberg, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States